CLINICAL TRIAL: NCT02674334
Title: Prospective Evaluation of Cognitive Outcomes After Anesthesia on Patients in the Beach Chair Position
Acronym: BCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, George K Bal, Associate Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1409418786
Record Dates: First submitted 2015-12-10; First posted 2016-02-04 (Estimated); Results first posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-08

CONDITIONS: Injury as a Result of Positioning
Keywords: orthopedic procedures
MeSH Terms: interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NIRS Monitored Not Treated (Active Comparator): Anesthesiologist blinded to Near Infrared Spectroscopy (NIRS)
  Interventions: Device: NIRS monitored not treated
- NIRS Monitored and Treated (Active Comparator): Anesthesiologist treats based on Near Infrared Spectroscopy (NIRS)
  Interventions: Device: NIRS

INTERVENTIONS:
Device: NIRS — Near infrared spectroscopy (NIRS) monitor allows anesthesiologist to treat cerebral desaturations according to NIRS results while maintaining Mean Arterial Pressure (MAP) at least 60mmHG or at least 80% of baseline
  Other Names: Near infrared spectroscopy
  Arms: NIRS Monitored and Treated
Device: NIRS monitored not treated — Near infrared spectroscopy (NIRS) monitored but anesthesiologist blinded to NIRS information and treatment is standard of care.
  Other Names: Near infrared spectroscopy
  Arms: NIRS Monitored Not Treated

SUMMARY:
The purpose of this study was to use Near Infrared Spectroscopy (NIRS) monitoring on participants undergoing shoulder surgery in the beach chair position (BCP) to determine cerebral desaturation events (CDE) and to further determine cognitive changes pre and post surgery using the Mini Mental State Exam.

DETAILED DESCRIPTION:
In this prospective, randomized, controlled study, investigators used a standardized anesthesia protocol to maintain the Mean Arterial Pressure (MAP) during surgeries done in the Beach Chair Position (BCP). Investigators hypothesized that, if the MAP was maintained, Near Infrared Spectroscopy (NIRS) monitoring would not change intra-operative anesthesia management and would not affect the post-operative cognitive outcomes of participants undergoing surgery in the beach chair position. Investigators secondarily wanted to document the actual incidence of cerebral desaturation events (CDEs) recorded by NIRS occurring in participants placed in the BCP if the MAP was strictly maintained.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* elective shoulder surgery in the beach chair position

Exclusion Criteria:

* less than 18 years of age
* preoperative score of 23 or less on the pre-operative Mini Mental State Exam
* traumatic brain injury
* transient ischemic attack
* cerebrovascular incident
* any apparent clinical neurologic dysfunction
* carotid artery stenosis
* known vascular malformation in head
* inability to have blood pressure measured in the opposite extremity
* malignant hyperthermia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George K Bal, MD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Only group data will be available.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were informed of the study in the Orthopaedic clinic at the visit prior to surgery. The consent form and pre- and post-testing using the Mini Mental State Examination (MMSE) was reviewed. Following consent, the baseline MMSE was administered. A score below 24 disqualified participants. Recruitment began October 2012 and ended May 2013.
Pre-assignment Details: Excluded reasons: anesthesiologist availability; surgery started early; illiteracy; less than 24 on the pre-operative MMSE; supine and BCP; no surgery; surgery delayed; operating suite could not accommodate NIRS monitor; data not recorded; previous difficult intubation; surgeon in two operating suites simultaneously; not needed, quota met.
Groups:
- NIRS Monitored Not Treated: Participants were monitored via near infrared spectroscopy (NIRS) for cerebral desaturation events during shoulder surgery in the beach chair position. Anesthesiologists were blinded to the NIRS data and treated participants based on standard of care treatment.
- NIRS Monitored and Treated: Participants were monitored via near infrared spectroscopy (NIRS) for cerebral desaturation events during shoulder surgery in the beach chair position. Anesthesiologists treated participants based on the NIRS monitoring in addition to standard of care.
Period: Overall Study
Arm/Group | NIRS Monitored Not Treated | NIRS Monitored and Treated
Started | 47 | 43
Completed | 40 | 40
Not Completed | 7 | 3
Not completed — Lost to Follow-up | 5 | 3
Not completed — participant difficulty breathing | 1 | 0
Not completed — NIRS not recording | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- NIRS Monitored Not Treated: Participants were monitored via near infrared spectroscopy (NIRS) for cerebral desaturation events during shoulder surgery in the beach chair position. Anesthesiologists were blinded to NIRS data and treated participants per standard of care.
- NIRS Monitored and Treated: Participants were monitored via near infrared spectroscopy (NIRS) for cerebral desaturation events during shoulder surgery in the beach chair position. Anesthesiologists treated participants based NIRS monitoring and per standard of care.
- Total: Total of all reporting groups
Arm/Group | NIRS Monitored Not Treated | NIRS Monitored and Treated | Total
Number analyzed (Participants) | 47 | 43 | 90
Age, Customized [Number; unit: participants] — >=18 years
  participants
    >=18 years | 47 | 43 | 90
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 31 | 29 | 60
Region of Enrollment [Number; unit: participants]
  United States | 47 | 43 | 90

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 20+% Cerebral Desaturation Events
Description: Cerebral desaturation event defined as a 20% or greater decrease from baseline Mean Arterial Pressure, while undergoing elective ambulatory surgery in the beach chair position
Time Frame: one day
Population: Participants undergoing elective shoulder surgery in the beach chair position at West Virginia University Medicine Hospital.
Measure: Count of Participants; unit: Participants
Groups:
- NIRS Monitored Not Treated: Participants were monitored via near infrared spectroscopy (NIRS) for cerebral desaturation events during shoulder surgery in the beach chair position. Anesthesiologists were blinded to the NIRS monitoring and treated participants per standard of care based on MAP.
- NIRS Monitored and Treated: Participants were monitored via near infrared spectroscopy (NIRS) for cerebral desaturation events during shoulder surgery in the beach chair position. Anesthesiologists treated participants based on NIRS monitoring results in addition to standard of care treatment based on MAP.
Arm/Group | NIRS Monitored Not Treated | NIRS Monitored and Treated
Number analyzed (Participants) | 40 | 40
Participants | 40 | 40

2. Secondary Outcome: Change in Mini Mental State Exam (MMSE) > 2 or a Score of 23 up to Two Weeks After Surgery Minus Baseline Value
Description: Change in total score of the MMSE measurement taken at baseline before surgery compared to the follow up measurement taken up to two weeks after surgery. Total range is zero to 30 with higher values indicating a better outcome. Indicator of cognitive decline measured by a change in Mini Mental State Exam (MMSE) > 2 or a score of 23 for two time points; up to two weeks after surgery minus the baseline value.
Time Frame: baseline and up to two weeks
Population: Participants who underwent elective shoulder surgery in the beach chair position at West Virginia University Medicine Hospital.
Measure: Mean (Standard Error); unit: scores on a scale
Units Other Than Participants: participants
Arm/Group | NIRS Monitored Not Treated | NIRS Monitored and Treated
Number analyzed (Participants) | 40 | 40
scores on a scale | -1.33 (.82) | -.17 (.16)
Statistical Analysis 1: Comparison: NIRS Monitored Not Treated vs NIRS Monitored and Treated; Test type: Superiority or Other; p = 0.165, ANOVA — P-values were not adjusted for multiple inferences; Continuous responses were tested using RCB ANOVA; Mean Difference (Net) = 1.16, 95% CI 2-sided [-.49 to 2.82], Standard Error of Mean 0.83

ADVERSE EVENTS:
Time Frame: 1 day
Description: Shoulder surgeries done as same-day surgery.
Arm/Group | NIRS Monitored Not Treated | NIRS Monitored and Treated
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/43
Other Adverse Events (participants affected / at risk) | 0/47 | 0/43

LIMITATIONS AND CAVEATS:
It is difficult to generalize the results of the study, few CDEs, to similar populations. Intubation may be related to the occurrence of CDEs or may have been related to patient co-morbidities and not the actual intubation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No